CLINICAL TRIAL: NCT06581484
Title: Improving Care for Adults With Congenital Heart Disease
Brief Title: Improving Congenital Heart Disease Care
Acronym: EmpowerMyCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: K23HL151866 (NIH); K23HL151866 (NIH)
Record Dates: First submitted 2024-08-19; First posted 2024-09-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Disease; Behavior, Health; Quality of Life; Empowerment, Patient; Activation, Patient
MeSH Terms: conditions — Heart Defects, Congenital; Health Behavior; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This is a digital (web and mobile-based) multicomponent patient engagement behavioral intervention. The intervention components include digital medical passport, health-specific updated information, credible resources, connections with the community, peer- and expert support and guidance, among others
  Interventions: Behavioral: Digital patient empowerment intervention

INTERVENTIONS:
Behavioral: Digital patient empowerment intervention — The intervention has features such as a digital medical passport, updated health-related information, community support and patient/peer stories and advice

SUMMARY:
The theory-informed digital health intervention, called as "Empower My Congenital Health (EmpowerMyCH)" aims to activate and engage ACHD patients in building confidence toward navigating the adult healthcare system. This tool is built after incorporating the theories of behavior change, gathering inputs from target patients in all stages of its design and implementation. The key features of the tool include a digital medical passport, updated congenital information, community support, and patient stories and advice. The investigators aim to test the acceptability, feasibility, efficacy, and effectiveness of the intervention.

DETAILED DESCRIPTION:
The goal of this clinical trial study is to learn whether a digital multi-component intervention would increase the knowledge, self-efficacy, self-advocacy, and patient engagement skills of adults with congenital heart disease (CHD) to confidently navigate the health care system and have timely recommended specialist visits.

The multicomponent intervention contains features such as a digital medical passport, updated health-related specific information, opportunities to engage with CHD community, peer-support, doctor visit reminders, etc. The intervention components are designed with inputs from the patients and the CHD community and have the potential to be adapted on an ongoing basis depending on the needs of the patients.

The main question it aims to answer is:

Does the digital multi-component CHD patient engagement intervention enhance the patient engagement skills and lead to timely specialist visit?

Participants will be recruited from the clinics, through word of mouth, social media, and others. Participants can use the website link or a QR code to sign an electronic consent form to be eligible to participate. Once consented, the participants will receive surveys to collect baseline and health status information as well as intervention components at regular intervals. The study will be available for participants to join on the web or mobile, depending on their preferences.

ELIGIBILITY:
Inclusion Criteria:

* have congenital heart disease
* 18 years or older
* can sign the informed consent

Exclusion Criteria:

* developmentally delayed
* unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 6-12 months
  Number of patients recruited out of all the eligible patient approached for recruitment
Satisfaction with the intervention components | 0, 6 and 12 months
  Scores on client satisfaction questionnaire (CSQ-8) survey. Scores are summed across items once. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Acceptability of the intervention components | 0, 6 and 12 months
  Rates of app downloads. The investigators will download app data monthly to evaluate the frequency and duration of the use of various intervention components.
  The investigators will recruit 10 participants for focused group discussions on acceptability of the app.
Feasibility of the intervention | 0, 6 and 12 months
  Ability to download the app or any technical difficulties with the app or its features.

SECONDARY OUTCOMES:
Patient activation measure (PAM) | 0, 6, 12 months
  The Patient Activation Measure® is a 13-item survey that assesses an individual's knowledge, skills and confidence integral to managing one's own health and healthcare. PAM generates a score along an empirical, interval-level scale from 0-100 that correlates to one of four levels of patient activation. PAM Levels 1 and 2 indicate lower patient activation, while PAM Levels 3 and 4 indicate higher patient activation.
Gothenburg Empowerment Scale (GES) | 0, 6, 12 months
  Each question is scored on a 5-point Likert scale, with 1 = strongly disagree and 5 = strongly agree. A higher total score indicates a higher level of empowerment.
  The GES is a validated and reliable measure of patient empowerment in adults with CHD. It can be used to assess empowerment levels over time, to identify areas where empowerment can be improved, and to evaluate the effectiveness of interventions to promote empowerment.
Timely specialist visit | 24 - 36 months
  Proportion with scheduled or completed ACHD specialist visits.
Euro-Quality of Life | 0, 6, 12, and 24 months
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. Higher score indicates worse quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Anushree Agarwal, MBBS, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No